CLINICAL TRIAL: NCT04660669
Title: Early Remote Intervention in Autism: a Randomized Noninferiority Clinical Trial Comparing Semi-intensive Early Start Denver Model (ESDM) Intervention With Remote Parental Training/ Supervision Versus Intensive ESDM Intervention.
Brief Title: Early Intervention in Remote Autism (IPAAD)
Acronym: IPAAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IPAAD (29BRC19.0279)
Record Dates: First submitted 2020-11-09; First posted 2020-12-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Early Intervention in Remote Autism
Keywords: Autism; ASD; ESDM; MOOC
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Group 1 receives 15 hours per week of ESDM intervention from ESDM therapists. The parents benefit from a 20 hour parent training program delivered in the participating center. Group 2 receives 8 hours per week of ESDM intervention from ESDM therapists in addition to whatever community service the parents choose. The parents benefit from a training program remotely delivered via a MOOC platform as well as parental supervision of sessions delivered at home 1 hour per week for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESDM 15h (Other): This arm receives 15 hours per week of ESDM intervention from ESDM therapists. The parents benefit from a 20 hour parent training program delivered in the participating center.
  Interventions: Other: ESDM intervention
- ESDM 8h + MOOC (Other): This arm receives 8 hours per week of ESDM intervention from ESDM therapists in addition to whatever community service the parents choose. The parents benefit from a training program remotely delivered via a MOOC platform as well as parental supervision of sessions delivered at home 1 hour per week for the duration of the study.
  Interventions: Other: ESDM intervention; Other: MOOC

INTERVENTIONS:
Other: ESDM intervention — Early Start Denver Model (ESDM) intervention with remote parental training/ supervision versus intensive ESDM intervention.
Other: MOOC — Massive Online Open Course: a teaching and learning intervention based on instrumental and interactive teaching situations
  Arms: ESDM 8h + MOOC

SUMMARY:
The Early Start Denver Model (ESDM) has shown its efficiency in the early management of ASD.

The study aims to evaluate the efficiency of a new type of management based on a semi-intensive center-based intervention (8h per week) coupled with a MOOC (Massive Online Open Course: a teaching and learning intervention based on instrumental and interactive teaching situations) for remote parental training/supervision. The goal is to determine if compared to the ESDM reference intervention (15h per week), this type of care can bring, a sufficient improvement in child development course and decreased symptoms of autism in young children, and if it could be, therefore, better suited to the needs of children and their family, bypassing the previously stated obstacles.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ASD based on the Diagnosis and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria;
2. Diagnosis of ASD on the Autism Diagnosis Observation Schedule (ADOS-2) and Autism Diagnosis Interview (ADIR) for toddlers (we will include children above or equal to 13, which is the research cut-off);
3. Aged between 15 and 36 months;
4. DQ of 30 or above at the MSEL
5. Sign informed consent form by both parents

Exclusion Criteria:

1. A neurodevelopmental disorder with known etiology (e.g. fragile X syndrome, Rett syndrom)
2. Significant sensory or motor impairment
3. Major physical problems such as a chronic serious health condition
4. History of a serious head injury and/or neurologic disease
5. Seizures at time of entry
6. Use of psychoactive medications (7 ) Families unavailable for the intervention and the followup over a period of 12 months

(8) Impossibility for family to have access to the MOOC

Ages: 15 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The gain in developmental quotient measured using the Mullen Scales of Early Learning (MSEL) | From day 0 to months 12
  Minimum = 49 (worse outcome) and maximum = 155 (better outcome)

SECONDARY OUTCOMES:
Assessment of child autism symptoms and change in autism symptoms using ADOS-2 | At baseline, 6 months after the set up of the intervention and at 12 months after the set up of the intervention
  Minimum = 0 (better outcome) and maximum = 28 (worse outcome)
Assessment of child behavioral adaptation using The Vineland Adaptive Behavior Scales second version (VABS-2) | At baseline, 6 months after the set up of the intervention and at 12 months after the set up of the intervention
  Minimum = 20 (worse outcome) and maximum = 160 (better outcome)
Assessment of sensory reactivity using The Dunn's Sensory Profile for toddlers | At baseline, 6 months after the set up of the intervention and at 12 months after the set up of the intervention
  Minimum = 38 (worse outcome) and maximum = 190 (better outcome)
Assessment of the parent burden and quality of life using the CareQuol-7D | At baseline, 6 months after the set up of the intervention and at 12 months after the set up of the intervention
  Minimum = 0 (worse outcome) and maximum = 100 (better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LAVENNE, Principal Investigator — CHRU BREST
Locations (4):
- France (4):
  - CH Réné-Dubos, Cergy-Pontoise
  - CHU Le Havre, Le Havre
  - CH Limoges, Limoges
  - CHU Nantes, Nantes